CLINICAL TRIAL: NCT04660006
Title: Optical Coherence Tomography Angiography Changes Post-cataract Surgery in Patients With and Without Diabetic Retinopathy
Brief Title: Diabetic Retinopathy and OCT-A Changes Post-cataract Surgery
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Uptown Eye Specialists (Other)
Responsible Party: Sponsor
Other Study IDs: OCTa Study 1.0
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Cataract; Diabetic Retinopathy; Macular Edema Due to Diabetes Mellitus
Keywords: Optical Coherence Tomography Angiography
MeSH Terms: conditions — Cataract; Diabetic Retinopathy | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: Patients undergoing uneventful cataract surgery with no retinal vascular disease.
  Interventions: Procedure: Cataract surgery
- Diabetic Retinopathy (DR): Patients with non-proliferative diabetic retinopathy with no diabetic macular edema treatment in the 6 months prior to uneventful cataract surgery.
  Interventions: Procedure: Cataract surgery
- Diabetic Macular Edema (DME): Patients with diabetic macular edema undergoing active Anti-VEGF treatment (within the last 3 months) undergoing uneventful cataract surgery.
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Procedure: Cataract surgery — Patients undergoing uneventful cataract surgery were recruited to this study if they met the inclusion criteria of the three groups. Postoperative retinal vasculature measures, as recorded by the optical coherence tomography angiography imaging technique, were compared to baseline measures.

SUMMARY:
The purpose of this study is to use optical coherence tomography angiography (OCT-A) to compare retinal vasculature after uncomplicated cataract surgery in patients with and without diabetic retinopathy.

DETAILED DESCRIPTION:
Patients undergoing cataract surgery who provided informed consent were enrolled in the study. There were three comparison groups: control, diabetic retinopathy (DR) and diabetic macular edema (DME) groups. Optical coherence tomography angiography (OCT-A) scans measuring retinal thickness, vessel density, perfusion density, and foveal avascular zone were obtained at baseline and postoperative week one, month one and month three.

ELIGIBILITY:
Inclusion Criteria:

* All patients at Uptown Eye Specialists undergoing uneventful cataract surgery who have provided informed consent to the study.

Exclusion Criteria:

* Other ocular co-morbidities such as axial length < 22.0 mm or > 25.0 mm, previous ocular surgeries, previous history of uveitis, previous ocular trauma, cornea pathologies or glaucoma, intraocular pressures over 22 mmHg
* In groups 1 and 2: previous retinal laser treatments
* OCT-A signal strength < 6
* Use of multifocal intraocular lens
* Second eye (if first eye recruited)
* In Group 1: No diabetes mellitus as past medical history

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants selected from Uptown Eye Specialists, an eye care clinic, at two sites in Brampton, Ontario, Canada and Vaughan, Ontario, Canada.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2019-05-27 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of retinal vessel density up to 3 months post-cataract surgery. | Preoperative (Baseline); Postoperative (1 Week, 1 Month, 3 Months)
  Optical coherence tomography angiography (OCT-A) scans will be taken at baseline and postoperative week one, month one, and month three. This imaging modality provides measurements for retinal vessel density to be compared between groups and time.
Change from baseline of retinal perfusion density up to 3 months post-cataract surgery. | Preoperative (Baseline); Postoperative (1 Week, 1 Month, 3 Months)
  Optical coherence tomography angiography (OCT-A) scans will be taken at baseline and postoperative week one, month one, and month three. This imaging modality provides measurements for retinal perfusion density to be compared between groups and time.
Change from baseline of foveal avascular zone up to 3 months post-cataract surgery. | Preoperative (Baseline); Postoperative (1 Week, 1 Month, 3 Months)
  Optical coherence tomography angiography (OCT-A) scans will be taken at baseline and postoperative week one, month one, and month three. This imaging modality provides measurements for foveal avascular zone (FAZ), particularly FAZ area, perimeter, and circularity index, to be compared between groups and time.
Change from baseline of retinal thickness up to 3 months post-cataract surgery. | Preoperative (Baseline); Postoperative (1 Week, 1 Month, 3 Months)
  Optical coherence tomography (OCT) scans will be taken at baseline and postoperative week one, month one, and month three. This imaging modality provides measurements of retinal thickness, particularly, central subfield and average macular cube thickness, to be compared between groups and time.

SECONDARY OUTCOMES:
Development of new cystoid macular edema | Preoperative (Baseline); Postoperative (1 Week, 1 Month, 3 Months)
  New cases of cystoid macular edema (a potential side effect of cataract surgery) are to be recorded to determine if there are preoperative risk factors for development of cystoid macular edema post-cataract surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah H Chiu, MD, FRCSC, Principal Investigator — Uptown Eye Specialists
Locations (1):
- Uptown Eye Speicialists, Brampton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eriksson U, Alm A, Bjarnhall G, Granstam E, Matsson AW. Macular edema and visual outcome following cataract surgery in patients with diabetic retinopathy and controls. Graefes Arch Clin Exp Ophthalmol. 2011 Mar;249(3):349-59. doi: 10.1007/s00417-010-1484-9. Epub 2010 Sep 9. PMID 20827486
- [Background] Yu S, Frueh BE, Steinmair D, Ebneter A, Wolf S, Zinkernagel MS, Munk MR. Cataract significantly influences quantitative measurements on swept-source optical coherence tomography angiography imaging. PLoS One. 2018 Oct 2;13(10):e0204501. doi: 10.1371/journal.pone.0204501. eCollection 2018. PMID 30278057
- [Background] Zhao Z, Wen W, Jiang C, Lu Y. Changes in macular vasculature after uncomplicated phacoemulsification surgery: Optical coherence tomography angiography study. J Cataract Refract Surg. 2018 Apr;44(4):453-458. doi: 10.1016/j.jcrs.2018.02.014. Epub 2018 Apr 25. PMID 29705010
- [Background] Sorour O, Arya M, Waheed N. New findings and challenges in OCT angiography for diabetic retinopathy. Annals of Eye Science. 2018; 3(8): 44-54.